CLINICAL TRIAL: NCT07054138
Title: Pre-operative Study the Efficacy of Nebulized Dexmedetomidine on Blunting Hemodynamic Changes During Intubation and Pneumoperitoneum in Morbid Obese Patients During Laparoscopic Bariatric Surgery: Randomized Double Blind Control Study
Brief Title: Efficacy of Nebulized Dexmedetomidine on Blunting Hemodynamic Changes During Intubation and Pneumoperitoneum in Morbid Obese Patients During Laparoscopic Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, AHMED ABDELAZIZ SHAMA, Assistant Professor of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KFSIRB200-20
Record Dates: First submitted 2025-06-03; First posted 2025-07-08 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Nebulization; Dexmedetomidine; Hemodynamic Changes; Intubation; Pneumoperitoneum; Morbid Obesity; Laparoscopic Bariatric Surgery
MeSH Terms: conditions — Pneumoperitoneum; Obesity, Morbid | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Experimental): Patients will be nebulized with dexmedetomidine 1 mcg/kg in 3 ml of 0.9 % saline 15 minutes before shifting the patients to the operating room with a face mask 6 L/min in a sitting position.
  Interventions: Drug: Dexmedetomidine
- Control group (Placebo Comparator): Patients will be nebulized with 3 ml of 0.9% normal saline 15 minutes before shifting the patients to operation room with face mask 6 L/min in sitting position.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Dexmedetomidine — Patients will be nebulized with dexmedetomidine 1 mcg/kg in 3 ml of 0.9 % saline 15 minutes before shifting the patients to the operating room with a face mask 6 L/min in a sitting position.
  Arms: Dexmedetomidine group
Drug: Normal Saline — Patients will be nebulized with 3 ml of 0.9% normal saline 15 minutes before shifting the patients to the operating room with a face mask, 6 L/min in a sitting position.
  Arms: Control group

SUMMARY:
This study aims to evaluate the effect of preoperative dexmedetomidine nebulization on blunting hemodynamic response for laryngoscope, intubation, pneumoperitoneum, and opioid consumption in morbidly obese patients undergoing laparoscopic bariatric surgery.

DETAILED DESCRIPTION:
Obesity is a major global public health issue. Morbidly obese patients have multiple pathophysiological changes that affect most of the body organs in the form of restrictive lung diseases, obstructive sleep apnea (OSA), hypertension, cardiovascular problems, metabolic syndrome, and fatty infiltration of the liver.

Direct laryngoscopy and intubation are noxious stimuli that are associated with transient, unpredictable, and variable hemodynamic changes. This response occurs within 30 seconds after intubation and lasts less than 10 minutes. The consequences of laryngoscopy and intubation may precipitate ischemia, arrhythmias, cerebrovascular stroke, pulmonary oedema, and an increase in the intracranial pressure in the vulnerable group.

Dexmedetomidine is an α2 adrenergic agonist that has been proven to attenuate the hemodynamic response to intubation and pneumoperitoneum, along with a dose-sparing effect on opioids and propofol. It has been used in multiple routes, including intravenous, intramuscular, oral, nasal, and intrathecal routes. Inhalation of the nebulized drug is non-invasive and associated with high bioavailability. Nebulized dexmedetomidine may offer an attractive alternative to both intravenous and intranasal routes of administration, as drug deposition following nebulization occurs over the nasal, buccal, and respiratory mucosa.

ELIGIBILITY:
Inclusion Criteria:

* Age from 20 to 60 years old.
* Both sexes.
* American Society of Anesthesiologists (ASA) Physical Status I-III.
* Morbidly obese patients with a body mass index (BMI) between 30 and 45.

Exclusion Criteria:

* Patients' refusal
* Decompansated hepatic, renal, or cardiac disease
* Expected difficult airway management
* Uncontrolled hypertension
* Psychiatric disease
* Sever pulmonary disease
* Patients on opioid, alcohol, beta-blockers, or allergy to any of the study drugs.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2025-07-10 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of increase in hemodynamic response | Intraoperatively
  Incidence of increase in hemodynamic response, either heart rate, mean arterial pressure, or both.

SECONDARY OUTCOMES:
Preoperative sedation score | Preoperatively
  Preoperative sedation score will be assessed using (Ramsay Sedation Scale): (1) Awake; agitated or restless or both, (2) Awake; cooperative, oriented and tranquil, (3) Awake but response to commands only,(4) Asleep; brisk response to light glabellar tab or loud auditory, (5) A sleep; sluggish response to light glabellar tab or loud auditory stimulus , (6) sleep; no response to glabellar tab or loud auditory stimulus.
Intraoperative fentanyl consumption | Intraoperatively
  Intraoperative fentanyl consumption will be recorded.
Intraoperative propofol consumption | Intraoperatively
  Intraoperative propofol consumption will be recorded.
Time for first use of rescue analgesia | 24 hours postoperatively
  Time for first use of rescue analgesia will be assessed from the end of surgery till first dose of morphine administrated.
Total opioid consumption | 24 hours postoperatively
  After assessment of pain scores, when numerical rating scale (NRS) measures more than 3; patients will receive 3mg morphine, which can be repeated considering that the total daily consumption of morphine never exceeds 20 mg.
Incidence of adverse effects | 24 hours postoperatively
  Incidence of adverse effects such as nausea, vomiting, bradycardia, hypotension or hypoxia will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.